CLINICAL TRIAL: NCT02883894
Title: Interest of Dosage of Anti-PB230, Anti-PB180 and Cytokines for Monitoring of Patients Suffering From Bullous Pemphigoid
Acronym: Cyto-PB
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 176IR09
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Blood Specimen Collection; Interleukin-17; Interleukin-23

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- bullous pemphigoid: Patients with bullous pemphigoid.
  Interventions: Other: Blood sample for dosages of cytokines (IL-17 and IL-23) and of the protease MMP-9

INTERVENTIONS:
Other: Blood sample for dosages of cytokines (IL-17 and IL-23) and of the protease MMP-9

SUMMARY:
Bullous pemphigoid is the most common subepidermal autoimmune blistering disease of the skin in European countries, including France.

Immunologically, BP is characterized by the production of autoantibodies directed against two major components of the hemidesmosome, BP180 and BP230.

The anti-BP180 autoantibody is detected in 79-93% of cases of bullous pemphigoid and its serum level at diagnosis have been correlated with disease activity. The anti-BP230 autoantibody is detected in 57%-63% of bullous pemphigoid cases and its score at diagnosis did not correlate with disease activity.

Up to now, no clinical or immunologic factors have been identified to predict outcome of patients with good or poor prognosis bullous pemphigoid as defined by long complete remission off therapy and recurrent disease requiring maintenance therapy for years. The usefulness of BP180 or BP230 ELISA scores for monitoring BP patients during treatment also remains unclear.

DETAILED DESCRIPTION:
Aim of the study were :

To study association between the serum level of cytokines (IL-17 and IL-23) and of the protease MMP-9 and the relapse of bullous pemphigoid.

ELIGIBILITY:
Inclusion Criteria:

* patients with bullous pemphigoid
* patients not yet receiving treatment for bullous pemphigoid
* aged > 18 years

Exclusion Criteria:

- Patients with relapse of bullous pemphigoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bullous pemphigoid.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Relapse of bullous pemphigoid. | Month 12
  The relapse of bullous pemphigoid is defined as he reappearance of at least 3 new daily blisters along with pruritus and/or erythematous, eczematous or urticarial plaques

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Plee J, Le Jan S, Giustiniani J, Barbe C, Joly P, Bedane C, Vabres P, Truchetet F, Aubin F, Antonicelli F, Bernard P. Integrating longitudinal serum IL-17 and IL-23 follow-up, along with autoantibodies variation, contributes to predict bullous pemphigoid outcome. Sci Rep. 2015 Dec 14;5:18001. doi: 10.1038/srep18001. PMID 26656739